CLINICAL TRIAL: NCT04476316
Title: Prevalence and Clinical Characterization of Traumatic Events in Women With Fibromyalgia
Brief Title: Prevalence of the Traumatic Events in Women With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Ana Moreno Alcázar, Principal Investigator, Parc de Salut Mar
Other Study IDs: 2020/9158
Record Dates: First submitted 2020-07-07; First posted 2020-07-20 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Fibromyalgia; Psychological Trauma; Pain; Anxiety; Depression; Sleep Disturbance; Quality of Life
MeSH Terms: conditions — Fibromyalgia; Psychological Trauma; Pain; Anxiety Disorders; Depression; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Suffering a traumatic event is a potential risk factor for developing Posttraumatic Stress Disorder (PTSD) with or without comorbidities with other pathologies that can become chronic with time, including fibromyalgia. Different study results show the existence of an association between living traumatic events and developing fibromyalgia. However, studies in the field have not evaluated thoroughly the nature of traumatic events, the subsequent development of PTSD and the degree to which it can cause an impairment. These results will allow us increase the knowledge about the effects of comorbidity between both medical conditions, get to know in depth the type of traumatic events that female patients with FM suffer, and express the importance of the implementation of a therapeutic approach which takes into account the existing psychological symptoms in addition to the main principal pathology.

DETAILED DESCRIPTION:
BACKGROUND:

Fibromyalgia (FM) affects 2-4% of the general population with typical symptoms being generalized and widespread pain, sleep disturbances, problems in memory and attention, anxiety and depression. Different studies have demonstrated a clear relationship between the presence of psychological trauma and FM, in terms of sexual and physical abuse, chronic stress and adverse lifetime events. According to some studies, the prevalence of Posttraumatic Stress Disorder (PTSD) in patients with FM is 45,3%, while in the general population it appears to be between 1.3%-12.3%. Nevertheless, current therapeutic approaches do not take into account the assessment and treatment of this risk factor, therefore the clinical benefits obtained are limited. Moreover, existing studies in the field do not carry out a thorough clinical characterization of these traumatic events. As a result, there is a lack of consensus about the prevalence of the different types of traumatic events and their temporality, as well as a lack of awareness of the level of interference and impairment in patients with FM. Additionally, studies done on the topic are subject to important methodological biases.

JUSTIFICATION OF THE STUDY:

Due to everything explained above, we consider that studying the prevalence and clinical characteristics of the possible traumatic events in patients with FM has a great relevance and clinical importance, due to the considerable negative impact they have across the beginning, curse and prognosis of this disease.

AIMS:

The main objective of the project is to study de prevalence and characterization of traumatic events in a sample of women diagnosed with FM and their association with FM's clinical severity.

Specifically, the study intends to analyze the existence of specific characteristics of traumatic events, such as the age when the event was experienced, the type of trauma (interpersonal o intrapersonal; simple or complex; single or repeated in time, etc.) that can be predictors or explicative of the patterns presented by these patients.

HYPOTHESIS:

1. Participants who have suffered traumatic events during childhood, of the interpersonal type and repeated in time will be associated with greater severity of FM and higher levels of pain.
2. Participants who have suffered traumatic events during childhood, of the interpersonal type and repeated in time will present greater severity in the clinical symptoms of trauma.
3. Participants who have suffered traumatic events during childhood, of the interpersonal type and repeated in time will present higher severity in affective symptoms, sleep disturbances and quality of life.

STUDY DESIGN:

This is a transversal descriptive study in which the Rheumatology Service, Adult Mental Health Service and Primary Care Centers of the Parc de Salut Mar will participate. The evaluations will be carried out in a single interview with the duration of 1 hour and a half, and will be conducted by specialized psychologists of the Centre Forum Research Unit (IMIM). Participants will have the choice to attend the assessment in the Centre Forum C/Llull 410, 08019) or in the Rheumatology Service (CAP Vila Olímpica, C/Joan Miró 17, 08005) of the Parc de Salut Mar.

During assessment sociodemographic, clinical and pharmacological data will be collected. Additionally, through the use of evaluation scales, pain and FM impact, psychological trauma related symptoms, clinical symptoms, insomnia and quality of life will be evaluated.

STATISTICAL ANALYSIS:

The data analysis will be carried out using the R statistics package. Logic, range and data consistency tests will be applied to clean the data. In the same way, the different distributions of the variables will be obtained in order to facilitate the detection of possible errors in the data entry.

Descriptive analysis will be carried out of all the identified variables in the study. Likewise, regression analysis will be used to predict the pain severity index (EVA, PDI, FIQ) based on trauma-related variables (CTQ, IES-R, SUD, DES, SDQ-20), and to predict the clinical severity index (HADS, AIS, SWLS) based on the pain-related variables (EVA, PDI, FIQ). Redundant variables will be eliminated from the model in order to identify the smallest possible group of predictors to explain a substantial amount of the variation in the dependent variables.

To control a possible confusion bias, an adjustment model will be defined to study the influence of other variables and analyse possible confounders.

A general lineal model will be used for independent variables of more than 2 categories and two sample t-tests will be used for variables of 2 categories. Where data does not meet criteria for parametric tests, non parametric tests will be used.

ELIGIBILITY:
Inclusion Criteria:

* Women with FM diagnosis.
* Age between 18-70.

Exclusion Criteria:

* Comorbid autoimmune or chronic inflammatory disease.
* Neurological or serious medical diseases.
* Severe mental health disorders such as bipolar disorder, schizoaffective disorder and/or schizophrenia.
* Active suicidal ideation.
* Substance abuse/dependence within 1 month prior to participation (except for nicotine abuse/dependency).

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study sample will consist in 83 patients diagnosed with FM recruited by different services of the Parc de Salut Mar.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Levels of pain assessed with the Visual Analogic Scale Questionnaire (VAS) | 1 week
  Severity in pain intensity will be assessed with the Visual Analogic Scale (rated in a continuum from 0 to 10).
Levels of pain assessed with the Pain Dissability Index (PDI) | 1 week
  Severity in pain intensity will be assessed with the Pain Disability Index (7 items rated from 0 to 10, making a total score from 0 to 70).
Levels of pain assessed with the Fibromyalgia Impact Questionnaire (FIQ) | 1 week
  Severity in pain intensity will be assessed with the Fibromyalgia Impact Questionnaire (the first items is rated from 0 to 4, the second from 0 to 7 and the third from 0 to 5; whereas the other 7 items are rated from 0 to 10, with a cut-off score of 50).
Presence of Postraumatic Stress Disorder (PTSD) evaluated with the Evaluación Global de Estrés Postraumático (EGEP-5) | 1 week
  Presence of Postraumatic Stress Disorder (PTSD) will be assessed using the EGEP-5, a 55-item clinician-administered scale based on DSM-V criteria. There are three different sections: presence of traumatic events, symptoms and functioning. The scale can determine a diagnosis of PTSD, specifying the presence of dissociative symptoms (depersonalization and derealization) and delayed expression.
Levels of trauma associated symptoms assessed with the Impact of Events Scale-Revised (IES-R) | 1 week
  Psychological trauma will be evaluated using the Impact of Events Scale-Revised. This scale consists in 22-item to determine frequency and impact of posttraumatic symptoms experienced, with subscales of intrusion, avoidance and hyperarousal, each scored on a 5-point Likert scale, yielding a score for each subscale and a total score. This scale has a scoring range of 0 to 88. On this test, scores that exceed 24 can be quite meaningful. High scores have the following associations: 24 or more PTSD is a clinical concern. Those with scores this high who do not have full PTSD will have partial PTSD or at least some of the symptoms; 33 and above represents the best cutoff for a probable diagnosis of PTSD; 37 or more this is high enough to suppress your immune system's functioning (even 10 years after an impact event).
Presence of stressful life events in the last year using Holmes & Rahe Social Readjustment Scale | 1 week
  This scale lists 43 possible stressful life events. Each of them have their respective scores. Global scores under 150 indicate low levels of stress, scores between 150 and 299 indicate a 50% risk of stress-related disorders and scores above 300 represent an 80% risk of suffering from stress.
Presence of childhood trauma assessed by Childhood Trauma Quiestionnaire (CTQ) | 1 week
  The CTQ is a self-administered scale which includes a 28-item test that measure 5 types of childhood maltreatment: emotional, physical and sexual abuse, and emotional or physical neglect. A 5-point Likert scale is used for the responses which range from never true to very often true (with total scores ranging from 5 to 25). The final scores provide a severity score for each subscale from "none to minimal," "low to moderate," "moderate to severe" and "severe to extreme".
Levels of dissociation evaluated by Dissociative Experiences Scale (DES) | 1 week
  The DES consists of 28 questions about different experiences related to dissociation, excluding when the subject has been under the effects of any substance. This test is scored by totaling the percentage answered for each question (from 0 to 100) and then dividing by 28. A total score higher than or equal to 30 corresponds with high levels of dissociation.
Levels of somatoform dissociation assessed by Somatoform Dissociation Questionnaire 20 (SDQ-20) | 1 week
  SDQ-20 is a 20-item self-report questionnaire measuring somatoform dissociation. Items refer to somatic symptoms and then ask if there is a known cause. The items are answered on a 5-point Likert scale and the symptoms with no known cause are summed to achieve the total score.
Levels of depressive symptoms assessed by with the Hospital Anxiety and Depression Scale (HADS) | 1 week
  Severity of depressive symptoms will be evaluated with the Hospital Anxiety and Depression Scale. Items are rated on a 4-point Likert scale from 0 and 3, yielding a total score ranging from 0 to 21 and a cut-off score of 8 indicating probable clinical symptoms.
Levels of anxious symptoms evaluated with the Hospital Anxiety and Depression Scale (HADS) | 1 week
  Severity of anxious symptoms will be evaluated with the Hospital Anxiety and Depression Scale. Items are rated on a 4-point Likert scale from 0 and 3, yielding a total score ranging from 0 to 21 and a cut-off score of 8 indicating probable clinical symptoms.
Presence of psyquiatric comorbid disorders assessed by MINI International Neuropsychiatric Interview | 1 week
  The MINI brief structured interview explores the principal psychiatric disorders from Axis I of DSM-IV and CIE-10. It is divided in different units and contains precise questions about the psychological problems which require yes/no answers.
Levels of sleep disturbances using Athens Insomnia Scale (AIS) | 1 week
  The AIS is a self-administered scale based on the ICD-10 criteria for insomnia. It measures sleep difficulties suffered over the previous three nights. It consists of 8 items evaluating sleep induction, awakenings during the night, final awakening, total sleep duration, sleep quality, well-being, functioning capacity and sleepiness during the day. It is scored from 0 to 24 and higher scores mean greater difficulties.
Levels of life satisfaction measured with Satisfaction With Life Questionnaire (SWLS) | 1 week
  The SWLS is a 5-item self-administered scale measuring global cognitive judgment of the satisfaction with one's life. The items can be rated from 1 to 5, and lower scores indicate lower satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Moreno-Alcázar, PhD., Principal Investigator — IMIM
Locations (1):
- Parc Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burke NN, Finn DP, McGuire BE, Roche M. Psychological stress in early life as a predisposing factor for the development of chronic pain: Clinical and preclinical evidence and neurobiological mechanisms. J Neurosci Res. 2017 Jun;95(6):1257-1270. doi: 10.1002/jnr.23802. Epub 2016 Jul 12. PMID 27402412
- [Background] Cabo-Meseguer A, Cerda-Olmedo G, Trillo-Mata JL. Fibromyalgia: Prevalence, epidemiologic profiles and economic costs. Med Clin (Barc). 2017 Nov 22;149(10):441-448. doi: 10.1016/j.medcli.2017.06.008. Epub 2017 Jul 19. English, Spanish. PMID 28734619
- [Background] Collado A, Gomez E, Coscolla R, Sunyol R, Sole E, Rivera J, Altarriba E, Carbonell J, Castells X. Work, family and social environment in patients with Fibromyalgia in Spain: an epidemiological study: EPIFFAC study. BMC Health Serv Res. 2014 Nov 11;14:513. doi: 10.1186/s12913-014-0513-5. PMID 25385047
- [Background] Hauser W, Galek A, Erbsloh-Moller B, Kollner V, Kuhn-Becker H, Langhorst J, Petermann F, Prothmann U, Winkelmann A, Schmutzer G, Brahler E, Glaesmer H. Posttraumatic stress disorder in fibromyalgia syndrome: prevalence, temporal relationship between posttraumatic stress and fibromyalgia symptoms, and impact on clinical outcome. Pain. 2013 Aug;154(8):1216-23. doi: 10.1016/j.pain.2013.03.034. Epub 2013 Apr 2. PMID 23685006
- [Background] Kok T, de Haan H, van der Meer M, Najavits L, de Jong C. Assessing traumatic experiences in screening for PTSD in substance use disorder patients: what is the gain in addition to PTSD symptoms? Psychiatry Res. 2015 Mar 30;226(1):328-32. doi: 10.1016/j.psychres.2015.01.014. Epub 2015 Jan 28. PMID 25687377
- [Background] Morgan B, Wooden S. Diagnosis and Treatment of Common Pain Syndromes and Disorders. Nurs Clin North Am. 2018 Sep;53(3):349-360. doi: 10.1016/j.cnur.2018.04.004. PMID 30100001
- [Background] Yavne Y, Amital D, Watad A, Tiosano S, Amital H. A systematic review of precipitating physical and psychological traumatic events in the development of fibromyalgia. Semin Arthritis Rheum. 2018 Aug;48(1):121-133. doi: 10.1016/j.semarthrit.2017.12.011. Epub 2018 Jan 10. PMID 29428291
- [Derived] Gardoki-Souto I, Redolar-Ripoll D, Fontana M, Hogg B, Castro MJ, Blanch JM, Ojeda F, Solanes A, Radua J, Valiente-Gomez A, Cirici R, Perez V, Amann BL, Moreno-Alcazar A. Prevalence and Characterization of Psychological Trauma in Patients with Fibromyalgia: A Cross-Sectional Study. Pain Res Manag. 2022 Nov 30;2022:2114451. doi: 10.1155/2022/2114451. eCollection 2022. PMID 36504759
- See also: Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences (2nd ed.). Hillsdale, NJ: Lawrence Erlbaum Associates, Publishers. — https://www.scirp.org/(S(lz5mqp453edsnp55rrgjct55))/reference/ReferencesPapers.aspx?ReferenceID=2041144
- See also: Martínez Ibáñez, J. J. (2010). Repensando el concepto de trauma. Una redefinición desde los aportes del psicoanálisis relacional. Clínica e Investigación Relacional, 4(3), 1-20. — https://www.psicoterapiarelacional.es/Portals/0/eJournalCeIR/V4N3_2010/04_JJMtnez-Iba%C2%A4ez_Repensando-Trauma_CeIR_V4N3.pdf?ver=2010-10-31-020500-000